CLINICAL TRIAL: NCT04513288
Title: ICITRU : Randomized Trial of Immunonutrition With L-citrulline in Patients Hospitalized in Intensive Care for Sepsis or Septic Shock
Acronym: ICITRU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC19_9778_ICITRU; 2020-A01804-35 (Other: ID RCB)
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, placebo-controlled, randomized, double-blind study on two parallel groups.
Who Masked: Participant
Masking Description: Prospective, multicenter, placebo-controlled, randomized, double-blind study on two parallel groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Enteral administration of citrulline for 5 days. L-citrulline (Protéocit®). This commercial form consists only of L-citrulline. Each patient will receive 10 grams per day in 2 doses (1 stick/ 12H = 5 grams / 12H). These sticks contain a powder to be resuspended in 50 mL of water for injection (ppi) for 1 stick. They will be delivered in a 50 mL syringe allowing administration of the product through the nasogastric tube. The solution will be prepared just before administration.
  Interventions: Dietary Supplement: Experimental treatment L-citrulline (Protéocit®)
- Control group (Placebo Comparator): Enteral administration of iso-nitrogenous placebo for 5 days. The placebo used will consist of a mixture of 4 non-essential amino acids. 5 g of L-citrulline provides 1.2 g of nitrogen. For the mixture to be iso-nitrogenous, each of the 4 amino acids will need to provide 0.3 g of nitrogen. The mixture will therefore consist of 21.6% alanine, 32.3% aspartate, 18.2% glycine and 27.9% proline for a total of 8.83 g of amino acids per sachet. 2 administrations (2 sticks) daily for 5 days.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Experimental treatment L-citrulline (Protéocit®) — Enteral administration of citrulline for 5 days.
  Arms: Experimental group
Other: Placebo treatment — Enteral administration of iso-nitrogenous placebo for 5 days.
  Arms: Control group

SUMMARY:
Immunonutrition in intensive care has not yet demonstrated a beneficial effect on organ failure, the acquisition of nosocomial infections, or mortality. It did not correct for acquired immunosuppression in intensive care patients. Despite numerous methodological problems (use of several pharmaconutrients, very heterogeneous set of patients) and the absence of clinical data, deleterious effects have been attributed to immunonutrition in intensive care, in particular in septic patients and patients in intensive care . Arginine (ARG) is a semi-essential amino acid involved in many immunological mechanisms. It is synthesized in sufficient quantity under normal conditions but quickly becomes insufficient under catabolic conditions such as in severe sepsis. Arginine is not only the precursor of nitrogen monoxide (NO) but also an essential substrate for numerous enzymatic reactions which participate in the maintenance of immune homeostasis, in particular T lymphocyte function. Depletion of the cellular medium in arginine will induce an abnormality in the metabolism of immune cells responsible for a dysfunction of these cells (lymphopenia linked to early apoptosis) and thus expose patients to organ failure and nosocomial infections.

It has been found that hypoargininemia in intensive care patients is associated with the persistence of organ dysfunction (SOFA score), the occurrence of nosocomial infections and mortality. Also, it has been demonstrated that in these patients, enteral administration of ARG was not deleterious and increased ornithine synthesis, suggesting a preferential use of ARG via the arginases route, without significant increase in argininaemia or effect on immune functions. L-citrulline (CIT), an endogenous precursor of ARG, constitutes an interesting alternative for increasing the availability of ARG. Sponsor recent data demonstrate that the administration of CIT in intensive care is not deleterious and that it very significantly reduces mortality in an animal model of sepsis, corrects hypoargininemia, with convincing data on immunological parameters such as lymphopenia, which is associated with mortality, organ dysfunction and the occurrence of nosocomial infections. The availability of ARG directly impacts the mitochondrial metabolism of T lymphocytes and their function. Our hypothesis is therefore that CIT supplementation is more effective than administration of ARG in correcting hypoargininemia, reducing lymphocyte dysfunction, correcting immunosuppression and organ dysfunction in septic patients admitted to intensive care.

DETAILED DESCRIPTION:
Strategy :

Enteral administration of citrulline for 5 days versus iso-nitrogenous placebo. Amino acid assay and immunological parameters (monocytic expression of HLA-DR, MDSCs, cytokines / chemokines, lymphocyte number and phenotype, apoptosis and lymphocyte proliferation and mitochondrial function and T lymphocyte repertoire) will only be carried out on patients included in Rennes (60 patients).

ELIGIBILITY:
Inclusion Criteria:

* Septic patients in accordance with the definition of sepsis and septic shock published in 2016 (JAMA) and whose use is recommended by the European Society of Intensive Care Medicine;
* Initial aggression dated less than 4 days before admission to intensive care (selection of "community" patients). The onset of aggression will be defined by the onset of clinical signs of infection;
* Patients hospitalized for less than 48 hours before admission to intensive care (selection of patients without malnutrition and immunosuppression acquired in hospital) *;
* Patients under invasive mechanical ventilation with a foreseeable ventilation duration> 2 days **;
* Exclusive enteral nutrition;
* Affiliation to a social security scheme;
* Consent signed by the patient, relative or legal representative or inclusion under emergency procedure

Non Inclusion Criteria:

* Progressive Sars-CoV2 infection
* Pregnancy in progress;
* Morbid obesity (BMI> 40);
* State of immunosuppression defined by at least one of these criteria: continuous administration of steroids at any dose for more than one month before hospitalization, steroids at high doses (> 0.5 mg / kg / day of methylprednisolone or equivalent), radiotherapy or chemotherapy in the previous year, proven humoral or cellular deficiency;
* Contraindication to enteral nutrition (SRLF 2016 recommendations: "Enteral nutrition should probably not be used upstream of a high flow digestive fistula in cases of intestinal obstruction, ischemia of the small intestine or digestive hemorrhage. active (Strong agreement) ");
* Participation in intervention research on a drug, or intervention research that could impact the immune system

Exclusion Criteria:

- Institution of immunosuppressive therapy such as chemotherapy, cyclophosphamide, high dose corticosteroid therapy (> 0.5 mg / kg / day ; hydrocortisone used in the management of septic shock is not considered an exclusion criterion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
SOFA score | Baseline and day 7 or last known SOFA score if the patient died or left intensive care before day 7.
  SOFA score for organ failure (5 parameters ranged from 0 to 4 each)

SECONDARY OUTCOMES:
Nosocomial infections | From Inclusion up to Day 28 maximum
  Incidence of nosocomial infections during the stay in intensive care (maximum Day 28). The diagnosis of nosocomial infections will be made by following the definitions of nosocomial infections of the CDC (Centers for Disease Control). An independent committee of experts will validate or not the infections.
Exposure to each antibiotic | Up to Day 28 maximum
  Number of days of exposure to each antibiotic per 1000 days of hospitalization (maximum Day 28)
Mortality in intensive care | Up to Day 28 maximum
  Mortality in intensive care
Hospital mortality | Up to Day 28 maximum
  Hospital mortality
Number and phenotypes of lymphocytes | Day 1, 3 and 7
  Number and phenotypes of lymphocytes on Day 1, Day 3 and Day 7
HLA-DR monocytic expression | Day 1, 3 and 7
  HLA-DR monocytic expression (flow cytometry) on Day 1, Day 3 and Day 7
Number of Myeloid-derived suppressor cells | Day 1, 3 and 7
  Number of Myeloid-derived suppressor cells (flow cytometry) at on Day 1, Day 3 and Day 7
Plasma cytokines / chemokines | Day 1, 3 and 7
  Plasma cytokines / chemokines (IL-6, IL-8, IL-10, IL-7, CXCL10, G-CSF, TNF-alpha, IFN-β) on on Day 1, Day 3 and Day 7
T repertoire | Day 1, 3 and 7
  Diversity of the T repertoire at Day 1, Day 3 and Day 7
T lymphocyte exhaustion | Day 1, 3 and 7
  T lymphocyte exhaustion: measurement of lymphocytic apoptosis and lymphocyte proliferation on Day 1, Day 3 and Day 7
Mitochondrial activity | Day 1, 3 and 7
  Measurement of mitochondrial activity (measurement of the number of mitochondria and their membrane potential, measurement of Beclin1 expression) on Day 1, Day 3 and Day 7
Plasma amino acids | Day 1, 3 and 7
  Plasma amino acids (arginine and its metabolites (ornithine, glutamate, glutamine, citrulline, proline) and tryptophan / kynurenine) on Day 1, Day 3 and Day 7
SOFA score | Day 3 and Day 5
  SOFA score for organ failures on Day 3 and Day 5 (5 parameters ranged from 0 to 4 each)
Duration of hospitalization in intensive care | Up to Day 28 maximum
  Duration of hospitalization in intensive care (days), up to Day 28 maximum
Duration of hospitalization at the hospital | Up to Day 28 maximum
  Hospital stay at the hospital (days), up to Day 28 maximum
Duration of mechanical ventilation | Up to Day 28 maximum
  Duration of mechanical ventilation (days), up to Day 28 maximum.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Rennes University Hospital - Medical ICU, Rennes, Brittany Region
  - Rennes University Hospital - Surgical ICU, Rennes, Brittany Region
  - Besançon University Hospital, Besançon
  - Le Mans Hospital, Le Mans
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided